CLINICAL TRIAL: NCT01132950
Title: Empowering Women to Make Contraceptive Choices While Incarcerated
Brief Title: Contraceptive Awareness and Reproductive Education
Acronym: CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial Hospital of Rhode Island (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Jennifer G. Clarke, MD, MPH, Memorial Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARE 07-42; 5R01HD054890 (NIH)
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Contraception; Sexually Transmitted Diseases; Pregnancy
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Didactic Educational Counseling (Active Comparator)
  Interventions: Other: Didactic Educational Counseling
- Motivation Interviewing (Experimental): Participant will receive two sessions of personalized motivational interviewing.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — Two personalized sessions of motivational interviewing. The first one is given while the participant is in jail and the second one is given at 3 months post release.
  Arms: Motivation Interviewing
Other: Didactic Educational Counseling — Participant will watch an educational video while in jail and a second educational video at 3 months post release.
  Arms: Didactic Educational Counseling

SUMMARY:
The purpose of this study is to increase the initiation and continuation of highly effective contraceptive use while incarcerated and upon release, as well as decrease unsafe sexual activity.

DETAILED DESCRIPTION:
Unplanned pregnancies and sexually transmitted infections are important and costly public health problems in the United States resulting from unprotected sexual activity. Women with a history of incarceration are at increased risk for these problems given the high rates of substance abuse and commercial sex work in this population. This proposal is designed to evaluate an innovative intervention Motivational Interviewing with Computer Assistance (MICA) designed to improve contraceptive use for incarcerated women who do not want a pregnancy and are soon to be released into the community. The investigators will utilize the Title X program which, in conjunction with RI Department of Corrections (RI DOC), provides reproductive health services in jail and then transitional services in the community after release. The investigators plan to recruit 400 women from the RI DOC women's jail and randomize them to two interventions: two sessions of personalized MICA or two sessions of Didactic Educational Counseling (DEC), both delivered individually by trained counselors. The two counseling interventions will be similar in length and timing, but will vary in content, counseling style and the individualized computer generated feedback that is reviewed with the counselor.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-35;
2. Currently sexually active with men defined as having coital sex at least monthly in the past three non-institutionalized months;
3. Expected place of residence after release in Providence County or within 15 miles of follow-up site;
4. Willing to comply with protocol, follow-up and provide at least one locator;
5. Fluent in English.

Exclusion Criteria:

1. Inability to give informed consent secondary to organic brain dysfunction, not having own legal guardianship, or active psychosis or otherwise not able to participate in the intervention or assessments (deaf, blind, or impaired communication skills that impair ability to participate in computerize assessment or counseling);
2. Pregnant or trying to become pregnant within the next year;
3. Hysterectomy, bilateral oophorectomy, tubal ligation, IUD or Essure (coil), implantable contraceptive devices (Implanon) or other procedures which make it very unlikely to become pregnant;
4. Women who are monogamous for more than one year whose partner has had a vasectomy;
5. Housed in segregation as we will be unable to recruit them for the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Contraceptive initiation | 5 years
  Initiation of a highly effective contraceptive method prior to release from jail will be limited to methods that are 98% or more effective in preventing pregnancy (Table 1).41 Initiation of these methods will be verified through review of the RI DOC medical records (as we have done in the past).
Continuous use of highly effective contraceptives at follow-up | 5 years
  If a participant switches from one highly effective contraceptive method to another she will be recorded as maintaining continuous contraceptive use at follow-up if she switches methods during times when the original method is still effective. Use of contraceptive methods will be confirmed through both TLFB and medical record review.
Incident STIs | 5 years
  At baseline participants will be tested for T. vaginalis, N. gonorrhoeae, and C. trachomatis through self obtained vaginal swabs. If a participant is diagnosed with an STI at baseline she will be treated and she will be asked to follow-up in six weeks for a test for cure. Any positive test after a baseline negative test will be documented as an incident infection.

SECONDARY OUTCOMES:
Incident pregnancy | 5 years
  An incident pregnancy will be defined as having occurred if there is a baseline negative pregnancy test and a positive urine Beta-HCG test through the study or a self reported pregnancy confirmed with a positive urine or serum Beta-hCG test through medical record review during the time of study participation. If a participant reports a positive pregnancy test outside of the study then she will be asked to sign a release of medical information form and a copy of the test results will be obtained.
Risk for unintended pregnancy and STIs | 5 years
  Risk behaviors will be determined through the TLFB. No or low risk for an unintended pregnancy will include either continuous use of a highly effective contraceptive method, abstinence, or use of a condom with a spermicide during every act of intercourse. No or low risk for STIs include abstinence or use of a condom with every act of intercourse and with every partner.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer G Clarke, MD, MPH, Principal Investigator — Memorial Hosptial of Rhode Island
Locations (1):
- Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States

REFERENCES:
- [Derived] Clarke J, Gold MA, Simon RE, Roberts MB, Stein L. Motivational interviewing with computer assistance as an intervention to empower women to make contraceptive choices while incarcerated: study protocol for randomized controlled trial. Trials. 2012 Jul 2;13:101. doi: 10.1186/1745-6215-13-101. PMID 22747705